CLINICAL TRIAL: NCT05281341
Title: Effect of Growth Hormone Administration With Controlled Ovarian Stimulation in Expected Poor Responders POSEIDON Group 3 and 4 Undergoing ICSI Using Antagonist Protocol
Brief Title: Effect of GH Administration in Poor Responders Undergoing Intracytoplasmic Sperm Injection (ICSI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305406
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-12

CONDITIONS: Female Infertility
Keywords: Growth hormone; Poor responder; Poseidon group,; ICSI
MeSH Terms: conditions — Infertility, Female | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poseidon Group 4A & 3A (Experimental): 80 eligible infertile women fulfilling the criteria of Poseidon Group 4 (35 years or more and AMH <1.2ng/ml) will be randomized into Group 4A will receive controlled ovarian stimulation (COS) and growth hormone (GH) and Group 4B will receive COS only. Similarly, 80 eligible infertile women fulfilling the criteria of Poseidon Group 3 (less than 35 years and AMH <1.2ng/ml) will be randomized into Group 3A will receive COS and GH and Group 3B will receive COS only.
  Interventions: Drug: Growth Hormone
- poseidon Group 4B & 3B (No Intervention): 80 eligible infertile women fulfilling the criteria of Poseidon Group 4 (35 years or more and AMH <1.2ng/ml) will be randomized into Group 4A will receive controlled ovarian stimulation (COS) and growth hormone (GH) and Group 4B will receive COS only. Similarly, 80 eligible infertile women fulfilling the criteria of Poseidon Group 3 (less than 35 years and AMH <1.2ng/ml) will be randomized into Group 3A will receive COS and GH and Group 3B will receive COS only.

INTERVENTIONS:
Drug: Growth Hormone — In GH groups (Group 4A & 3A), patients will receive additional treatment with GH (Somatropin, 4 IU/day, subcutaneous injection), daily beginning on the initial day of gonadotropin stimulation until triggering the oocyte maturation by hCG. Control groups (Group 4B & 3B) will receive only standard COS without GH supplementation
  Other Names: somatropin 4 IU
  Arms: Poseidon Group 4A & 3A

SUMMARY:
Despite the use of various treatment strategies, poor response to ovarian stimulation remains a major clinical challenge with lower chance to obtain sufficient number of oocytes and thus less likely to conceive with high risk of cycle cancellation. The aim of this study is to evaluate the effect of recombinant human GH administration to gonadotropins on clinical and laboratory ICSI outcomes in expected poor responders more and less than 35 years (Poseidon group 4 and 3 respectively).

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women aged 20-45 years.
2. AFC <5.
3. AMH level <1.2 ng/ml.
4. Have two normal ovaries and normal uterine cavity.

Exclusion Criteria:

1. Body mass index (BMI) >30 kg/m2.
2. Follicle Stimulating Hormone (FSH) > 15 IU/L.
3. History of abnormal karyotype in one or both partners.
4. Endocrine, metabolic or autoimmune disorders, such as diabetes, thyroid disorder, and polycystic ovary syndrome (PCOS).
5. Women with a known medical disease (e.g. severe hypertension or hepatic disease).
6. Endometriosis.
7. Previous ovarian surgery.
8. Current or history of malignancies, chemotherapy or radiotherapy.
9. Severe male actor (total motile sperm count <1×106 or normal morphology <1%)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-02-13 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 28 gestational weeks
  calculated as the number of live births (defined as at least one live born after 28 weeks of gestation) divided by the total number of patients who performed pregnancy tests.

SECONDARY OUTCOMES:
Serum E2 level | 2-3 weeks
  Serum Estradiol level on day of human chorionic gonadotropin (hCG) in pg.
Endometrial thickness | 2-3 weeks
  Endometrial thickness on day of hCG in mm
Fertilization rate | 1 day after oocyte retrieval
  number of 2pn oocytes to the total number of injected oocytes
Number of day 3 embryos | 3 days after oocyte retrieval
  Total number of available embryos on day 3 after oocyte retrieval
Clinical pregnancy rate | 2 weeks after positive pregnancy test
  Calculated as the number of clinical pregnancies (defined as the presence of a gestational sac with positive heart beat detected by transvaginal ultrasound scan 2 weeks after positive pregnancy test) divided by the number of embryo transfer procedures
Implantation rate | 2 weeks after positive pregnancy test
  Calculated as the ratio of the number of gestational sacs detected by sonography to the total number of embryos transferred
Miscarriage rate | 20 weeks
  The number fetal losses per clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Anis, phD, Principal Investigator — Alexandria University
Locations (1):
- faculty of medicine, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Oudendijk JF, Yarde F, Eijkemans MJ, Broekmans FJ, Broer SL. The poor responder in IVF: is the prognosis always poor?: a systematic review. Hum Reprod Update. 2012 Jan-Feb;18(1):1-11. doi: 10.1093/humupd/dmr037. Epub 2011 Oct 10. PMID 21987525
- [Background] Abu-Musa A, Haahr T, Humaidan P. Novel Physiology and Definition of Poor Ovarian Response; Clinical Recommendations. Int J Mol Sci. 2020 Mar 19;21(6):2110. doi: 10.3390/ijms21062110. PMID 32204404
- [Background] Humaidan P, Alviggi C, Fischer R, Esteves SC. The novel POSEIDON stratification of 'Low prognosis patients in Assisted Reproductive Technology' and its proposed marker of successful outcome. F1000Res. 2016 Dec 23;5:2911. doi: 10.12688/f1000research.10382.1. eCollection 2016. PMID 28232864
- [Background] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Background] Xu YM, Hao GM, Gao BL. Application of Growth Hormone in in vitro Fertilization. Front Endocrinol (Lausanne). 2019 Jul 23;10:502. doi: 10.3389/fendo.2019.00502. eCollection 2019. PMID 31396161
- [Background] Li XL, Wang L, Lv F, Huang XM, Wang LP, Pan Y, Zhang XM. The influence of different growth hormone addition protocols to poor ovarian responders on clinical outcomes in controlled ovary stimulation cycles: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Mar;96(12):e6443. doi: 10.1097/MD.0000000000006443. PMID 28328856
- [Background] Yang P, Wu R, Zhang H. The effect of growth hormone supplementation in poor ovarian responders undergoing IVF or ICSI: a meta-analysis of randomized controlled trials. Reprod Biol Endocrinol. 2020 Jul 29;18(1):76. doi: 10.1186/s12958-020-00632-w. PMID 32727608